CLINICAL TRIAL: NCT02815423
Title: Safety and Exploratory Efficacy Study of UCMSCs in Patients With Fracture and Bone Nonunion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Collaborators: Guangzhou Panyu Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-6
Record Dates: First submitted 2016-04-20; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-03

CONDITIONS: Fracture; Bone Nonunion
MeSH Terms: conditions — Fractures, Bone | interventions — Administration, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSCs (Experimental): Transplantation of umbilical cord mesenchymal stem cells (UCMSCs) in patients with fracture and bone nonunion.
  Interventions: Biological: UCMSCs
- Placebo (Placebo Comparator): The patients with fracture and bone nonunion who underwent percutaneous injection of placebo.
  Interventions: Biological: Percutaneous

INTERVENTIONS:
Biological: UCMSCs — Transplatation of umbilical cord mesenchymal stem cells
  Arms: UCMSCs
Biological: Percutaneous — Percutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of the present study is to evaluate the safety and exploratory efficacy of the umbilical cord mesenchymal stem cells for patients with fracture and bone nonunion.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with non union in the site of bone fracture and nonunion.
* Age more than 18 and less than 60 years old.
* Nonunion or delayed union.

Exclusion Criteria:

* Diagnosis of cancer.
* Pregnancy or breastfeeding.
* Patient positive by serology or PCR for HIV, hepatitis B or C infection the patient with Accompanied fracture such as hip fracture that could not weight bearing.
* Any medical or psychiatric condition that in the researcher´s opinion could affect the patient´s ability to complete the trial or hamper the participation in the trial.
* Patients do not sign the consent forms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Radiological progression of bone fusion | 12 months
  After patients receiving mesenchymal stem cells or placebo, imaging control by X-ray and CT, and then analysis by software(ImageJ ) at 1, 6 and 12 months

SECONDARY OUTCOMES:
Comparison of the rate of complications between the 2 groups | 12 months
Incidence of increased temperature sensitivity by questionnaire | 6 months
Incidence and severity of infections at grafting sites by questionnaire | 6 months

IPD SHARING:
Plan to Share IPD: Yes